CLINICAL TRIAL: NCT07173621
Title: Comparing the Impact of AMNIOEFFECT Application vs Standard of Care on Post-Operative Healing in Patients Who Have Undergone Thyroid and Parathyroid Surgery Via the Transcutaneous Approach
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sarasota Memorial Health Care System (Other)
Collaborators: MiMedx Group, Inc. (Industry)
Responsible Party: Principal Investigator, Ralph Tufano, Principal Investigator, Sarasota Memorial Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-SURG-34
Record Dates: First submitted 2025-09-07; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Thyroid; Wound; Parathyroid Diseases; Surgical Incision; Incision
Keywords: thyroid; parathyroid; surgery
MeSH Terms: conditions — Thyroid Diseases; Wounds and Injuries; Parathyroid Diseases; Surgical Wound

STUDY DESIGN:
Intervention Model Description: During the study, 334 patients who are to undergo transcutaneous thyroid or parathyroid surgery will be recruited to participate over a one-year period. A sample size of approximately 300 patients (150 per group), assuming a drop-out rate of 10%, a total sample size of 334 will be enrolled. Using a randomized control approach, the study would be conducted to evaluate the impact of AMNIOEFFECT placed over the strap muscle closure before the subcutaneous tissues and skin are reapproximated, compared to standard of care on post-operative pain, swallowing ability, and cosmesis (conferring of beauty) as indicated by scar appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amnioeffect Application (Experimental): AMNIOEFFECT placed over the strap muscle closure before the subcutaneous tissues and skin are reapproximated.
  Interventions: Other: Amnioeffect
- No Amnioeffect Application (No Intervention): No AMNIOEFFECT placed over the strap muscle closure before the subcutaneous tissues and skin are reapproximated

INTERVENTIONS:
Other: Amnioeffect — Amnioeffect is a placental-based allograft made of lyophilized human amnion/intermediate/chorion membrane (LHACM)
  Arms: Amnioeffect Application

SUMMARY:
The purpose of this study is to understand how placing Amnioeffect on patients having transcutaneous thyroid or parathyroid surgery affects surgery scar appearance, pain, and the ability to swallow and compare it to patients who do not have anything placed during surgery. The Food and Drug Administration regulates the use of Amnioeffect for homologous use. Both Amnioeffect application and no Amnioeffect application are considered standard of care; however, for the purpose of this study, the use of Amnioeffect during surgery will be considered the intervention, and no Amnioeffect application will be the standard of care.

DETAILED DESCRIPTION:
A product called AMNIOEFFECT has been developed as a barrier intended for use in the treatment of acute and chronic wounds, providing a protective environment to support the healing process. Manufactured by the company MIMEDX, it is a placental-based allograft made of lyophilized human amnion/intermediate/chorion membrane (LHACM). During the study, 334 patients who are to undergo transcutaneous thyroid or parathyroid surgery will be recruited to participate over a one-year period. Using a randomized control approach, the study would be conducted to evaluate the impact of AMNIOEFFECT placed over the strap muscle closure before the subcutaneous tissues and skin are reapproximated, compared to standard of care on post-operative pain, swallowing ability, and cosmesis (conferring of beauty) as indicated by scar appearance.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Patients undergoing thyroid/parathyroid surgery via a transcutaneous incision
* Participants must be willing and able to consent and take part in the study

Exclusion Criteria:

* Patients < 18 years old
* Pregnant patients
* Patients with a history of keloid scarring
* Patients who refuse blood products
* Previous neck surgery
* Patients on immunosuppressive medications (steroids, immune modulators, etc.)
* Patients with a known sensitivity to aminoglycoside antibiotics
* Patients with an active or latent infection
* Patients with a disorder that would create an unacceptable risk of post-operative complications
* Subjects may be excluded at the discretion of the physician(s) based on their clinical judgment and/or if the health or safety of the participant may be potentially impacted by taking part in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2027-10-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of scar appearance | Pre-procedure, 1 month post procedure, 3 months post procedure
  Measured by use of the Vancouver Scar Scale; scores rating on vascularity, pigmentation, pliability, and height. Total score ranges from 0-13, with 0 being "normal" appearance.
Determine swallowing effectiveness | Pre-procedure, 1 month post procedure, 3 months post procedure
  Measured by use of the SWAL-QOL score; this survey uses a Likert scale rating to ask questions regarding swallowing difficulties and associated quality of life impacts. Higher scores reflect lower impact on quality of life; lower scores would indicate higher impact.
Improvement in Pain Score | Pre-procedure, 1 month post procedure, 3 months post procedure
  Measured by use of the Visual Analog Scale; scoring 0 for no pain-10 for unbearable pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Sarasota Memorial Health Care System, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yilmaz S, Habibi HA, Yildiz A, Altunbas H. Thyroid Embolization for Nonsurgical Treatment of Nodular Goiter: A Single-Center Experience in 56 Consecutive Patients. J Vasc Interv Radiol. 2021 Oct;32(10):1449-1456. doi: 10.1016/j.jvir.2021.06.025. Epub 2021 Jul 10. PMID 34256121
- [Background] Watt T, Cramon P, Hegedus L, Bjorner JB, Bonnema SJ, Rasmussen AK, Feldt-Rasmussen U, Groenvold M. The thyroid-related quality of life measure ThyPRO has good responsiveness and ability to detect relevant treatment effects. J Clin Endocrinol Metab. 2014 Oct;99(10):3708-17. doi: 10.1210/jc.2014-1322. Epub 2014 Jul 8. PMID 25004246
- [Background] Sonbol HS. Extracellular Matrix Remodeling in Human Disease. J Microsc Ultrastruct. 2018 Jul-Sep;6(3):123-128. doi: 10.4103/JMAU.JMAU_4_18. PMID 30221137
- [Background] Koob TJ, Lim JJ, Zabek N, Massee M. Cytokines in single layer amnion allografts compared to multilayer amnion/chorion allografts for wound healing. J Biomed Mater Res B Appl Biomater. 2015 Jul;103(5):1133-40. doi: 10.1002/jbm.b.33265. Epub 2014 Aug 30. PMID 25176107
- [Background] Joshi CJ, Hassan A, Carabano M, Galiano RD. Up-to-date role of the dehydrated human amnion/chorion membrane (AMNIOFIX) for wound healing. Expert Opin Biol Ther. 2020 Oct;20(10):1125-1131. doi: 10.1080/14712598.2020.1787979. Epub 2020 Jul 20. PMID 32580594
- [Background] Dean DS, Gharib H. Epidemiology of thyroid nodules. Best Pract Res Clin Endocrinol Metab. 2008 Dec;22(6):901-11. doi: 10.1016/j.beem.2008.09.019. PMID 19041821
- [Background] Cheng KL, Liang KW, Lee HL, Wang HY, Shen CY. Thyroid artery embolization of large solitary symptomatic benign thyroid nodules through transradial approach. Quant Imaging Med Surg. 2023 Aug 1;13(8):5355-5361. doi: 10.21037/qims-22-1385. Epub 2023 May 30. PMID 37581037
- See also: AMNIOEFFECT PRODUCT BROCHURE — https://www.mimedx.com/wp-content/uploads/2023/11/US-LS-2100002-v2.0-AMNIOEFFECT-PRODUCT-BROCHURE-vF.pdf
- See also: AMNIOEFFECT Application Guide — https://www.mimedx.com/wp-content/uploads/2023/11/US-LS-2200005-v1.0_AMNIOEFFECT-Application-Guide.pdf
- See also: Processing — https://www.mimedx.com/processing/
- See also: Spine and Neurosurgery — https://www.mimedx.com/spine-and-neurosurgery/